CLINICAL TRIAL: NCT05219565
Title: Phase III, Open-label, Community-based, Cluster Randomised Controlled Trial to Evaluate the Efficacy, Cost-effectiveness, and Acceptability of Attractive Targeted Sugar Baits (ATSB) for Malaria Burden Reduction in Western Kenya
Brief Title: Evaluating ATSBs for Malaria Reduction in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); PATH (Other); Kenya Ministry of Health (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-027
Record Dates: First submitted 2021-08-02; First posted 2022-02-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2023-08

CONDITIONS: Malaria
Keywords: ATSB; Malaria; Kenya
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: Using restricted randomization criteria, eighty clusters will be randomized 1:1 to either the intervention arm (ATSBs deployed throughout the cluster) or the control arm. The clusters will be followed in parallel for two years. In year one the first and second cohort were enrolled and followed up over 6 months each. In year 2, the third cohort was enrolled and followed up over 1 year.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attractive Targeted Sugar Bait (ATSB) (Experimental): Clusters within the ATSB arm will have 2 ATSBs hung on all eligible structures in the cluster where consent from the corresponding compound has been given.
  Interventions: Device: Attractive Targeted Sugar Bait (ATSB)
- Control (No Intervention): Clusters within the control arm will not receive ATSBs.

INTERVENTIONS:
Device: Attractive Targeted Sugar Bait (ATSB) — An ATSB is a A4-sized panel containing thickened fruit syrup laced with a neonicotinoid insecticide, dinotefuran. The syrup-insecticide mixture is covered with a protective membrane that allows mosquitoes to feed through the membrane while preventing non-target organisms from feeding. This device is designed to attract and kill mosquitoes.
  Other Names: Attractive Toxic Sugar Bait
  Arms: Attractive Targeted Sugar Bait (ATSB)

SUMMARY:
The effectiveness of long-lasting insecticidal nets (LLINs) and indoor residual spraying (IRS) in western Kenya are threatened by insecticide resistance and vector behaviour changes toward early evening and outdoor biting malaria vectors. New tools to control malaria are needed to reduce and even interrupt malaria transmission. Attractive Targeted Sugar Bait (ATSB) is a promising new intervention designed to attract and kill mosquitoes, including those that IRS and LLINs do not effectively target. The ATSB 'bait stations' are A4-sized panels containing thickened fruit syrup laced with a neonicotinoid insecticide, dinotefuran, to attract and kill the foraging vectors. Entomological field trials in western Mali showed that ATSBs successfully reduce mosquito densities and longevity and thus have the potential to reduce malaria transmission. In Kenya, the investigators will conduct an open-label cluster-randomized controlled trial in 80 village clusters (40 per arm) to evaluate the effect of ATSBs on the burden of malaria. During two years, households in half of these village clusters will receive two or three ATSB bait stations per household structure on exterior walls approximately 1.8 meters above the ground. ATSBs will be replaced every six months. The primary outcome will be the incidence of clinical malaria in children aged 1-<15 years enrolled in a prospective cohort followed monthly for about six months each during a 2-year period. Secondary outcomes include malaria infection prevalence assessed by rapid diagnostic tests through household surveys and the case burden of clinical malaria assessed by passive facility-based and community-based surveillance. The study includes entomological monitoring and nested acceptability, feasibility, and health economics studies. The stand-alone trial in western Kenya is a part of a multi-country ATSB consortium conducting similar trials in Zambia and Mali.

DETAILED DESCRIPTION:
The current malaria vector control tools, long-lasting insecticidal nets (LLINs) and indoor residual spraying (IRS) are critically important and have saved many lives. However, their effectiveness in western Kenya is threatened by insecticide resistance and vector behaviour changes toward more early evening and outdoor biting malaria vectors. LLINs and IRS specifically target indoor-biting and indoor-resting mosquitoes. Malaria vectors exhibit different behavioural characteristics that mitigate the effectiveness of vector control strategies. For example, traditionally, An. gambiae s.s. has been regarded as human-biting with late-night indoor-feeding and indoor-resting behaviours, while An. Arabiensis is found more often in drier environments and is more zoophagic with outdoor biting and resting behaviours. Following LLINs and IRS's widespread scale-up, the dominant African vectors' distributions and behaviours changed with An. gambiae s.s. and An. Funestus (also an indoor human biter) diminishing in abundance relative to An. arabiensis. Subsequently, shifts towards earlier evening biting by An. Gambiae s.s. (before people enter houses to sleep under LLINs) and later biting by An. Funestus (biting in the morning after sunrise) are examples of behavioural plasticity enabling these species to avoid contact with the LLIN and IRS insecticides.

There is a need for interventions that supplement and complement LLINs and IRS by killing mosquitoes outside houses using other biologic mechanisms (e.g., targeting sugar feeding behaviour). Furthermore, insecticides are required with novel modes of action that may restore sensitivity to pyrethroids by killing both pyrethroid-resistant and sensitive mosquitoes. Attractive Targeted Sugar Bait (ATSB) (the name was recently changed from Attractive Toxic Sugar Bait to highlight that it targets malaria vectors) is a promising new intervention that potentially fills the need for outdoor interventions with novel killing effects.

ATSB 'bait stations' are A4-sized panels containing thickened fruit syrup laced with a neonicotinoid insecticide (dinotefuran) to attract and kill the foraging vectors. Entomological field trials in Mali showed that ATSBs successfully reduce mosquito densities and longevity and thus have the potential to reduce malaria transmission. Large scale efficacy studies are now needed to establish the efficacy of ATSB for controlling malaria transmission.

ELIGIBILITY:
Eligibility criteria for clusters: Inclusion criteria

* A grouping of contiguous rural villages in Alego-Usonga and Rarieda sub-counties of Siaya County
* A minimum of 200 households

Eligibility criteria for clusters: Exclusion criteria

* Hard to reach in the rainy season
* Refusal to participate by village elders

Eligibility criteria for participants in the cohort study: Inclusion criteria

* A resident of a household within the core area of a study cluster, defined as living in the household in the recent four months and planning to live in the same household for the next 6.5 months
* Aged ≥ 1 year and < 15 years at the time of enrollment
* Written informed consent and/or assent

Eligibility criteria for participants in the cohort study: Exclusion criteria

* A confirmed or suspected pregnancy. Pregnant women are excluded because they are eligible for intermittent preventive treatment of malaria in pregnancy (IPTp).
* Taking daily cotrimoxazole prophylaxis (because this has antimalarial effects)
* Known sickle cell disease (because they received antimalarial prophylaxis)
* Contraindication to artemether-lumefantrine, the medication used for parasite clearance

Eligibility criteria for households for ATSB deployment: Inclusion criteria

--Households located within one of the 40 clusters (core or buffer area) randomly allocated to the trial intervention arm with a least one permanent resident

Eligibility criteria for households for ATSB deployment: Exclusion criteria

* Refusal of consent by the head-of-household to deploy ATSB on the outer walls (intervention villages only)
* Vacated compounds

Eligibility criteria for households for entomological monitoring: Inclusion criteria

* Household located within the core area of the cluster
* Head of household or his/her representative is at least 18 years of age
* Written informed consent for the collection of entomological data by the head of household or representative

Eligibility criteria for households for entomological monitoring: Exclusion criteria --No residents sleeping in the household during the planned night of monitoring

Eligibility criteria for human landing catches: Inclusion criteria

* Men aged 18 to 49 years
* Willingness and ability to work late at night for up to 7 hours at a time
* Willingness to take and tolerate a treatment regimen of the appropriate Kenya Ministry of Health (MoH) recommended antimalarial and chemoprophylaxis with 250 mg of mefloquine weekly to prevent malaria starting two weeks before the start of and until four weeks after completing HLCs
* Written informed consent

Eligibility criteria for human landing catches: Exclusion criteria

* Refusal/inability to work late at night for up to 7 hours at a time
* Unwillingness to take or intolerance/allergy to appropriate MoH treatment regimen or chemoprophylaxis

Eligibility criteria for participants in rapid ethnographic methods evaluation (community members): Inclusion criteria

* A resident of a household within an intervention area defined as an ATSB area during the main trial or an ASB area during any preliminary studies
* Resides in a household at the time of ASB/ATSB deployment, where the ASB/ATSB was installed for at least one month.
* 18 years of age or older if participating in focus group discussions; 15 years of age or older if participating in in-depth interviews

Eligibility criteria for participants in rapid ethnographic methods evaluation (community members): Exclusion criteria

--Unable to provide consent

Eligibility criteria for participants in rapid ethnographic methods evaluation (ATSB monitoring assistants): Inclusion criteria

* Inclusion criteria ethnographic evaluation (ATSB monitoring assistants)
* Serving as an ATSB monitoring assistant with experience installing ATSBs and monitoring the deployment Eighteen years of age or older

Eligibility criteria for participants in rapid ethnographic methods evaluation (ATSB monitoring assistants): Exclusion criteria

* Less than one month experience (i.e. is new to the job)
* Unable to provide consent

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2962 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Clinical malaria | Two years
  The incidence rate of clinical malaria defined as current fever (axillary temperature of ≥37.5°C) or history of fever in last 48 hours and a positive rapid diagnostic test (RDT, pLDH or HRP2), in children aged 1-<15 years enrolled in the cohort study

SECONDARY OUTCOMES:
Time to first malaria infection by PCR | Two years
  The time to first malaria infection assessed by PCR in children aged 1-<15 years enrolled in a cohort study
Malaria infection incidence by RDT (pLDH) | Two years
  The incidence rate of malaria infection detected by RDT (pLDH) in children aged 1-<15 years enrolled in a cohort study
Malaria infection prevalence by RDT (pLDH) | Two years
  The prevalence of malaria infection detected by RDT (pLDH) in cross-sectional household surveys
Incidence of malaria illness (passive surveillance) | Two years
  The incidence rate of malaria illness (sick-visit with a positive malaria rapid diagnostic test or microscopy) assessed by health-facility and community-based surveillance
Incidence of non-malaria illness (cohort) | Two years
  The incidence rate of non-malaria illness in children aged 1-<15 years enrolled in a cohort study
Incidence of non-malaria illness (passive surveillance) | Two years
  The incidence rate of non-malaria illness assessed by health-facility and community-based surveillance
Prevalence of non-malaria illness | Two years
  The prevalence of non-malaria illness in cross-sectional household surveys
Malaria vector density | Two years
  Entomological outcome: Malaria vector densities
Proportion of female anopheles mosquitoes older than three gonotrophic cycles, | Two years
  Entomological outcome: The proportion of female anopheles mosquitoes older than three gonotrophic cycles.
Sporozoite rate | Two years
  Entomological outcomes: Sporozoite rate
Entomological Inoculation Rate (EIR) | Two years
  Entomological outcome: Entomological Inoculation Rate (EIR)
Non-Target Organisms (NTOs) attracted to ATSBs | Two years
  Entomological outcome: Proportion of monitoring visits where NTOs were observed on bait stations
Markers of insecticide resistance (dinotefuran) | Two years
  Entomological outcome: Proportion of mosquitoes with resistance to dinotefuran among total mosquitoes collected in 4 WHO mosquito tubes in the trial area
Markers of insecticide resistance (permethrin) | Two years
  Entomological outcome: Proportion of mosquitoes with resistance to permethrin among total mosquitoes collected in 4 WHO mosquito tubes in the trial area
Markers of insecticide resistance (deltamethrin) | Two years
  Entomological outcome: Proportion of mosquitoes with resistance to deltamethrin among total mosquitoes collected in 4 WHO mosquito tubes in the trial area
Antibody concentrations against malaria antigen MSP-1 | Two years
  Antibody concentration against merozoite surface protein-1 (MSP-1) among cohort participants
Antibody concentrations against malaria antigen CSP | Two years
  Antibody concentration against circumsporozoite proteins (CSP) among cohort participants
Complexity of infection (COI) | Two years
  The complexity of (malaria) infection assessed by molecular markers, including, but not limited to, 24-single-nucleotide polymorphisms (24-SNP) barcodes
Mosquito salivary antigens | Two years
  Presence of mosquito salivary antigens in human blood as a measure for mosquito biting rates among cohort participants
AEs | Two years
  Number of adverse events associated with misuse of ATSBs.
ATSB removal rate | Two years
  The proportion of ATSBs that have been moved/removed
Perceptions of ATSBs | Two years
  The proportion of household heads who perceive ATSBs as safe and effective out of all household head who consented to ATSB deployment on their household structures.
Household use of LLINs in the setting of ATSBs | Two years
  The proportion of children aged 1-<15 years enrolled in a cohort study who used an LLIN the night prior
Household care seeking behavior in the setting of ATSBs | Two years
  The proportion of children aged 1-<15 years enrolled in a cohort study who sought care for febrile illness
Cost-effectiveness | Two years
  Incremental cost-effectiveness of ATSB above the standard of care measured through costing of intervention and efficacy outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Samuels, MD, MHS, Principal Investigator — Centers for Disease Control and Prevention; Eric Ochomo, Principal Investigator — Kenya Medical Research Institute
Locations (9):
- Kenya (9):
  - Naya Health Centre, Siaya, Siaya County
  - Benga Dispensary, Siaya, Siaya County
  - Boro Dispensary, Siaya, Siaya County
  - Manyuanda Health Centre, Siaya, Siaya County
  - Nyadhi Dispensary, Siaya, Siaya County
  - Ong'ielo Model Health Centre, Siaya, Siaya County
  - Rabar Dispensary, Siaya, Siaya County
  - Rageng'ni Dispensary, Siaya, Siaya County
  - Rambugu Dispensary, Siaya, Siaya County

IPD SHARING:
Plan to Share IPD: Yes
The full protocol will be available on request to any interested professional and may be published in a peer-reviewed journal or deposited in an online repository. Individual, de-identified participant data will be made available for meta-analyses as soon as the data analysis is completed, with the understanding that the meta-analysis results will not be published before the individual trial results without the prior agreement of the investigators. The de-identified data set of the complete participant-level data will be available for sharing purposes, such as via the WWARN repository platform (http://www.wwarn.org/working-together/sharing-data/accessing-data). A Data Access Committee will consider all requests for data for secondary analysis to ensure that the use of data is within the terms of consent and ethics approval.
Supporting Information: Study Protocol, SAP
Time Frame: The full protocol and SAP will be published within the next 2 years. The individual de-identified data when data analysis is completed, within 6 months of trial completion.
Access Criteria: A Data Access Committee will consider all requests for data for secondary analysis to ensure that the use of data is within the terms of consent and ethics approval.

REFERENCES:
- [Background] Huho B, Briet O, Seyoum A, Sikaala C, Bayoh N, Gimnig J, Okumu F, Diallo D, Abdulla S, Smith T, Killeen G. Consistently high estimates for the proportion of human exposure to malaria vector populations occurring indoors in rural Africa. Int J Epidemiol. 2013 Feb;42(1):235-47. doi: 10.1093/ije/dys214. Epub 2013 Feb 9. PMID 23396849
- [Background] Amek N, Bayoh N, Hamel M, Lindblade KA, Gimnig JE, Odhiambo F, Laserson KF, Slutsker L, Smith T, Vounatsou P. Spatial and temporal dynamics of malaria transmission in rural Western Kenya. Parasit Vectors. 2012 Apr 28;5:86. doi: 10.1186/1756-3305-5-86. PMID 22541138
- [Background] Moiroux N, Damien GB, Egrot M, Djenontin A, Chandre F, Corbel V, Killeen GF, Pennetier C. Human exposure to early morning Anopheles funestus biting behavior and personal protection provided by long-lasting insecticidal nets. PLoS One. 2014 Aug 12;9(8):e104967. doi: 10.1371/journal.pone.0104967. eCollection 2014. PMID 25115830
- [Background] Sougoufara S, Diedhiou SM, Doucoure S, Diagne N, Sembene PM, Harry M, Trape JF, Sokhna C, Ndiath MO. Biting by Anopheles funestus in broad daylight after use of long-lasting insecticidal nets: a new challenge to malaria elimination. Malar J. 2014 Mar 28;13:125. doi: 10.1186/1475-2875-13-125. PMID 24678587
- [Background] Killeen GF. Characterizing, controlling and eliminating residual malaria transmission. Malar J. 2014 Aug 23;13:330. doi: 10.1186/1475-2875-13-330. PMID 25149656
- [Background] Killeen GF, Marshall JM, Kiware SS, South AB, Tusting LS, Chaki PP, Govella NJ. Measuring, manipulating and exploiting behaviours of adult mosquitoes to optimise malaria vector control impact. BMJ Glob Health. 2017 Apr 26;2(2):e000212. doi: 10.1136/bmjgh-2016-000212. eCollection 2017. PMID 28589023
- [Background] Zhu L, Muller GC, Marshall JM, Arheart KL, Qualls WA, Hlaing WM, Schlein Y, Traore SF, Doumbia S, Beier JC. Is outdoor vector control needed for malaria elimination? An individual-based modelling study. Malar J. 2017 Jul 3;16(1):266. doi: 10.1186/s12936-017-1920-y. PMID 28673298
- [Background] Traore MM, Junnila A, Traore SF, Doumbia S, Revay EE, Kravchenko VD, Schlein Y, Arheart KL, Gergely P, Xue RD, Hausmann A, Beck R, Prozorov A, Diarra RA, Kone AS, Majambere S, Bradley J, Vontas J, Beier JC, Muller GC. Large-scale field trial of attractive toxic sugar baits (ATSB) for the control of malaria vector mosquitoes in Mali, West Africa. Malar J. 2020 Feb 14;19(1):72. doi: 10.1186/s12936-020-3132-0. PMID 32059671
- [Background] Beier JC, Muller GC, Gu W, Arheart KL, Schlein Y. Attractive toxic sugar bait (ATSB) methods decimate populations of Anopheles malaria vectors in arid environments regardless of the local availability of favoured sugar-source blossoms. Malar J. 2012 Feb 1;11:31. doi: 10.1186/1475-2875-11-31. PMID 22297155
- [Background] Fiorenzano JM, Koehler PG, Xue RD. Attractive Toxic Sugar Bait (ATSB) For Control of Mosquitoes and Its Impact on Non-Target Organisms: A Review. Int J Environ Res Public Health. 2017 Apr 10;14(4):398. doi: 10.3390/ijerph14040398. PMID 28394284
- [Background] Marshall JM, White MT, Ghani AC, Schlein Y, Muller GC, Beier JC. Quantifying the mosquito's sweet tooth: modelling the effectiveness of attractive toxic sugar baits (ATSB) for malaria vector control. Malar J. 2013 Aug 23;12:291. doi: 10.1186/1475-2875-12-291. PMID 23968494
- [Background] Pocock SJ. When (not) to stop a clinical trial for benefit. JAMA. 2005 Nov 2;294(17):2228-30. doi: 10.1001/jama.294.17.2228. No abstract available. PMID 16264167
- [Background] Protopopoff N, Mosha JF, Lukole E, Charlwood JD, Wright A, Mwalimu CD, Manjurano A, Mosha FW, Kisinza W, Kleinschmidt I, Rowland M. Effectiveness of a long-lasting piperonyl butoxide-treated insecticidal net and indoor residual spray interventions, separately and together, against malaria transmitted by pyrethroid-resistant mosquitoes: a cluster, randomised controlled, two-by-two factorial design trial. Lancet. 2018 Apr 21;391(10130):1577-1588. doi: 10.1016/S0140-6736(18)30427-6. Epub 2018 Apr 11. PMID 29655496
- [Background] Gimnig JE, Walker ED, Otieno P, Kosgei J, Olang G, Ombok M, Williamson J, Marwanga D, Abong'o D, Desai M, Kariuki S, Hamel MJ, Lobo NF, Vulule J, Bayoh MN. Incidence of malaria among mosquito collectors conducting human landing catches in western Kenya. Am J Trop Med Hyg. 2013 Feb;88(2):301-8. doi: 10.4269/ajtmh.2012.12-0209. Epub 2012 Dec 18. PMID 23249685
- [Derived] Ogwang C, Samuels AM, McDermott DP, Kamau A, Lesosky M, Obiet K, Janssen JM, Odongo W, Gimnig JE, Gutman JR, Schultz JS, Towett O, Seda B, Chepkirui M, Muchoki M, Omondi S, Kosgei J, Polo B, Aduwo F, Otieno K, Donnelly MJ, Kariuki S, Ochomo E, Kuile FT, Staedke SG. Attractive targeted sugar baits for malaria control in western Kenya (ATSB-Kenya) - Effect of ATSBs on epidemiologic and entomologic indicators: A Phase III, open-label, cluster-randomised, controlled trial. PLOS Glob Public Health. 2025 Jun 26;5(6):e0004230. doi: 10.1371/journal.pgph.0004230. eCollection 2025. PMID 40570028
- [Derived] Kamau A, Obiet K, Ogwang C, McDermott DP, Lesosky M, Janssen J, Odongo W, Gutman JR, Schultz JS, Nicholas W, Seda B, Chepkirui M, Aduwo F, Towett O, Otieno K, Donnelly MJ, Ochomo E, Kariuki S, Samuels AM, O Ter Kuile F, Staedke SG. Attractive targeted sugar baits for malaria control in western Kenya (ATSB-Kenya): enrolment characteristics of cohort children and households. Malar J. 2024 Dec 30;23(1):403. doi: 10.1186/s12936-024-05234-0. PMID 39736740
- [Derived] Attractive Targeted Sugar Bait Phase III Trial Group. Attractive targeted sugar bait phase III trials in Kenya, Mali, and Zambia. Trials. 2022 Aug 9;23(1):640. doi: 10.1186/s13063-022-06555-8. PMID 35945599

DOCUMENTS (2):
  • Study Protocol (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/65/NCT05219565/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT05219565/SAP_001.pdf